CLINICAL TRIAL: NCT01942434
Title: The Influence of FADS2 rs 174575 on Breastmilk Fatty Acid Levels and the Recognition Memory Abilities of 6-month Old Breastfed Infants and Follow-up
Brief Title: Fatty Acid Levels and Memory in Breastfed Children
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Carol Cheatham, PhD, Assistant Professor of Psychology, University of North Carolina, Chapel Hill
Other Study IDs: 09-1869
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Cognitive Development
Keywords: Fatty acids; Breast milk nutrients; Cognitive development; Electrophysiology; Long-term assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To explore the relation between breastmilk nutrients and the cognitive abilities of breastfed infants.

Phase 1: Near 3 months of age child and mother saliva samples for DNA obtained with breast milk sample.

Phase 2: At 6 months of age child participates in electrophysiology session to test recognition memory.

Phase 3: At 26 or 38 months of age, children will complete behavioral, dietary, and physical assessments.

ELIGIBILITY:
Inclusion Criteria:

* typically-developing
* exclusively breastfed
* unremarkable delivery

Exclusion Criteria:

* non-English speaking
* history of seizure activity

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Breastfeeding infants and their mothers
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Relation between recognition memory and maternal FADS genotype | 6 months
  At 6 months of age, during the second session (Phase 2)

SECONDARY OUTCOMES:
Nutrient content of breastmilk as it relates to FADS genotype | 3 to 4 months
  Sample provided in session 1 when the infant was 3-4 months old (Phase 1)
Nutrient content of breastmilk as it relates to recognition memory | 6 months
  At 6 months of age, during the second session (Phase 2)
Relation between declarative memory and breastmilk nutrients | 26 or 38 months
  At session 3, when the child was either 26 or 38 months of age (Phase 3)
Relation between declarative memory and concurrent nutrients | 26 or 38 months
  At session 3, when the child was either 26 or 38 months of age (Phase 3)

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, PhD, Principal Investigator — UNC at Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States